CLINICAL TRIAL: NCT02885207
Title: Interest Balance Auto-immune Population in Patients With Focal Epilepsy of Unknown Cause, Not Structural, Not Genetics, Newly Diagnosed
Acronym: IBADEPIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00785-42
Record Dates: First submitted 2014-10-09; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Epilepsy
Keywords: Limbic encephalitis; anti-neuronal antibodies
MeSH Terms: conditions — Epilepsy; Limbic Encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal epilepsy of unknown cause (Other)
  Interventions: Biological: Focal epilepsy of unknown cause

INTERVENTIONS:
Biological: Focal epilepsy of unknown cause — Male or female 18-65 years presenting focal epilepsy on the following arguments:
  * Crisis with clinical symptoms indicating focal seizure
  * & / Or crisis or critical focal inter-recorded EEG interpreted by a neurologist with expertise in the field of epilepsy.
  From unknown cause:
  * No evidence of injury (excluding temporal or hyperintensity of hippocampal sclerosis) on brain MRI with focus on regions of interest cuts.
  * No discharge or generalized photosensitivity recorded over an extended interpreted by a neurologist with expertise in the field of epilepsy video-EEG.
  * No argument for metabolic or neurodegenerative genetic epilepsy.
  * Normal neurological examination. Epilepsy that started within a maximum period of 2 years prior to inclusion in the study (including vegetative symptoms of temporal focal seizures).
  Without treatment by benzodiazepines or anti-epileptics first-line monotherapy (excluding benzodiazepines).

SUMMARY:
The knowledge of encephalitis associated with antibodies targeting intracellular antigens, and neuronal surface antibody syndromes has expanded considerably in recent times.

The primary purpose of the investigators protocole is to determine the incidence of anti-neuronal antibodies (blood and CSF) in a population of patients suffering from focal epilepsy of unknown cause to guide the management of these patients.

The investigators hypothesis is that dysimmune encephalitis is more common than is suggested by the current literature, and that sometimes forms of encephalitis dysimmune "at minimum" can be observed only in the form of focal epilepsy without further manifestation associated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years
* Presenting focal epilepsy on the following arguments

  * Crisis with clinical symptoms indicating focal seizure
  * & / Or crisis or critical focal inter-recorded on EEG interpreted by a neurologist with expertise in the field of epilepsy.
* Having not yet received a CSF analysis
* From unknown cause:

  * No evidence of injury (excluding temporal or hyperintensity of hippocampal sclerosis) on brain MRI with focus on regions of interest cuts.
  * No discharge or generalized photosensitivity recorded over an extended interpreted by a neurologist with expertise in the field of epilepsy video-EEG.
  * No argument for metabolic or neurodegenerative genetic epilepsy.
  * Normal neurological examination.
* Epilepsy that started within a period of two years preceding the study entry (including vegetative symptoms of temporal focal seizures).
* Without treatment or as benzodiazepines or taking anti-epileptic first-line monotherapy (excluding benzodiazepines).
* Informed consent signed
* affiliated with a social security scheme

Exclusion Criteria:

* structural abnormality found in brain MRI (except temporal hyperintensity and / or sclerosis of the hippocampus).
* Background Neurological: hyperthermic seizures in childhood, neonatal distress, history of seizures related to a circumstance, inflammation or infection of the CNS.
* Taking toxic: chronic alcoholism, narcotic consumption
* The case for a genetic / metabolic neurodeg ear /: generalized EEG / photosensitivity / family history of epilepsy / autism / disorder syndrome psychomotor development / dysmorphic syndrome / extrapyramidal syndrome associated discharge
* History of thyroiditis or m. system (LEAD, SGS, PR, Sarcoidosis)
* Immunosuppression innate or acquired
* IC lumbar puncture or have already received a lumbar puncture before inclusion in the protocol.
* Person under supervision or guardianship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
anti-neuronal antibodies | 2 years
  Incidence of seropositive patients for anti-neuronal antibodies in a cohort of patients with focal epilepsy of unknown cause.

SECONDARY OUTCOMES:
statistically significant differences between people with and without-neuronal antibodies differences | 2 years
  Related to population characteristics: age, sex, ethnicity, handedness, immune dysfunction associated field, psychiatric field associated migraine associated

OTHER OUTCOMES:
Serum analysis:(composite measure) | 2 years
  Directed by a blood test on a peripheral vein: ANA, anti-ENA, anti-DNA, ANCA, anti-TPO, anti-TGO, APL, anti-GAD, anti-transglutaminase / anti-Hu, Yo, Ri, CV2 , amphiphysin, Ma2 / VGKC complex, anti-NMDA-R, anti-AMPA-R, anti-GABA B-R / Other: NFS, CRP, ESR, TSH, PT, APTT
CSF analysis (composite measure) | 2 years
  A lumbar puncture is performed under strict aseptic conditions, in the absence cons classic indications (abnormal crushes or platelet count) in hospital, followed by monitoring at least three hours, looking for: ac neurons anti / Finding an oligoclonal distribution (DOC, immunoglobulin synthesis intrathéquale) / WBC and red blood cells, protein level

CONTACTS AND LOCATIONS:
Overall Officials: BENOILID Aurélien, MD, Principal Investigator — not affiliated
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - CHU de Dijon, Dijon
  - CHU de Nancy, Nancy
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No